CLINICAL TRIAL: NCT07367087
Title: A Prospective Intra-Patient Randomized Controlled Trial Comparing Silver Sulfadiazine Combined With Hyaluronic Acid Versus Silver Sulfadiazine Alone in Bilateral Partial-Thickness Burns
Brief Title: Silver Sulfadiazine With Hyaluronic Acid Versus Silver Sulfadiazine Alone in Partial-Thickness Burns
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Muhammad Naveed Shahzad (Other)
Responsible Party: Sponsor-Investigator, Dr Muhammad Naveed Shahzad, Assistant Professor of Plastic Surgery, Nishtar Medical University
Organization: Nishtar Medical University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SSDHA-PTB-2026
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Partial-Thickness Burn, Thermal Burn
MeSH Terms: interventions — Silver Sulfadiazine; Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Intra-patient randomized controlled design in which each participant receives both interventions applied to bilateral burn wounds.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silver Sulfadiazine Plus Hyaluronic Acid (Experimental): Intra-patient burn areas treated with topical silver sulfadiazine combined with hyaluronic acid.
  Interventions: Drug: Silver Sulfadiazine With Hyaluronic Acid
- Silver Sulfadiazine Alone (Active Comparator): Intra-patient burn areas treated with topical silver sulfadiazine alone.
  Interventions: Drug: Silver Sulfadiazine

INTERVENTIONS:
Drug: Silver Sulfadiazine With Hyaluronic Acid — Topical application of silver sulfadiazine combined with hyaluronic acid applied once daily until complete re-epithelialization.
  Arms: Silver Sulfadiazine Plus Hyaluronic Acid
Drug: Silver Sulfadiazine — Topical application of silver sulfadiazine applied once daily until complete re-epithelialization.
  Arms: Silver Sulfadiazine Alone

SUMMARY:
Partial-thickness burns are commonly treated with topical silver sulfadiazine; however, its use may delay epithelialization due to cytotoxic effects on regenerating cells. Hyaluronic acid has biological properties that may enhance wound healing when combined with silver sulfadiazine. This study aims to compare the time to re-epithelialization between silver sulfadiazine combined with hyaluronic acid and silver sulfadiazine alone in patients with bilateral partial-thickness burns using an intra-patient randomized controlled design.

DETAILED DESCRIPTION:
This is a prospective, intra-patient randomized controlled clinical trial conducted at a tertiary care burn center. Patients of all ages presenting with bilateral, symmetrical partial-thickness thermal burns will be enrolled, provided the burn areas are clinically comparable and suitable for intra-patient randomized treatment.

In each patient, one burn area will be randomly assigned to receive topical silver sulfadiazine combined with hyaluronic acid, while the contralateral burn area will receive silver sulfadiazine alone.

Randomization will be performed at the wound level so that each participant serves as their own control, minimizing inter-individual variability. Both interventions will be applied using identical dressing techniques and schedules. The primary outcome measure is time to re-epithelialization, defined as the number of days from initiation of treatment to achievement of complete epithelial coverage of the wound surface.

Participants will be monitored daily until epithelialization is complete. This study is designed to evaluate whether the addition of hyaluronic acid to standard silver sulfadiazine therapy accelerates wound healing in partial-thickness burns under routine clinical conditions.

ELIGIBILITY:
Inclusion Criteria

Patients with acute bilateral partial-thickness (second-degree) thermal burns where both sides/areas are comparable and suitable for intra-patient treatment (one area treated with SSD+HA and the contralateral area with SSD alone)

Presentation within 72 hours of burn injury

Small to moderate total burn surface area suitable for conservative topical management

Burn wounds not requiring immediate excision or grafting at baseline

Ability to comply with daily dressing application and follow-up until complete re-epithelialization

Written informed consent from patient; for minors, parent/guardian consent and assent where applicable

Exclusion Criteria

Full-thickness (third-degree) burns or mixed-depth burns in the study areas

Chemical, electrical, radiation, or inhalational burns requiring ICU or ventilatory support

Infected burn wounds at baseline requiring systemic antibiotics

Major comorbidities likely to impair wound healing (e.g., uncontrolled diabetes, severe peripheral vascular disease, immunosuppression, severe malnutrition)

Known hypersensitivity to silver sulfadiazine, sulfonamides, hyaluronic acid, or formulation components

Pregnancy or lactation (as per institutional policy)

Non-comparable bilateral burn wounds

Concurrent participation in another interventional wound or burn study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Time to Complete Re-epithelialization | Up to 21 days
  Time (in days) from initiation of topical treatment to complete re-epithelialization of the partial-thickness burn wound, defined as full epithelial cover without exudate.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad N Shahzad, MBBS, MCPS,FCPS,FCPS, Principal Investigator — Department of Plastic Surgery, Nishtar Medical University / Nishtar Hospital Multan
Locations (1):
- Nishtar Medical University & Hospital, Multan, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No